CLINICAL TRIAL: NCT01710722
Title: The Effect of Leptin A-200, Caffeine/Ephedrine and Their Combination Upon Weight Loss and Body Composition in Man
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 20034
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — caffeine, ephedrine drug combination; lepa protein, zebrafish; Caffeine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- caffeine and ephedrine (Experimental): Caffeine 200 mg tablets and ephedrine HCl 25 mg tablets three times a day with placebo leptin A-200 subcutaneously once daily.
  Interventions: Drug: caffeine and ephedrine
- leptin A (Experimental): Leptin A-200 20 mg subcutaneously once daily and placebo tablets of caffeine and ephedrine three times a day.
  Interventions: Drug: Leptin A
- caffeine, ephedrine, and leptin A (Experimental): Caffeine 200 mg tablets and ephedrine HCl tablets 25 mg three times a day with leptin A-200 20 mg subcutaneously once daily.
  Interventions: Drug: caffeine, ephedrine, and leptin A

INTERVENTIONS:
Drug: caffeine and ephedrine — Caffeine 200 mg tablets and ephedrine HCl 25 mg tablets three times a day with placebo leptin A-200 subcutaneously once daily.
  Arms: caffeine and ephedrine
Drug: Leptin A — Leptin A-200 20 mg subcutaneously once daily and placebo tablets of caffeine and ephedrine three times a day.
  Arms: leptin A
Drug: caffeine, ephedrine, and leptin A — Caffeine 200 mg tablets and ephedrine HCl tablets 25 mg three times a day with leptin A-200 20 mg subcutaneously once daily.
  Arms: caffeine, ephedrine, and leptin A

SUMMARY:
The purpose of this study is to compare three treatments to see which causes the most weight loss, fat loss, loss of stomach fat and improvement in blood tests like cholesterol.

DETAILED DESCRIPTION:
Three treatments are compared to see which causes the most weight loss, fat loss, loss of stomach fat and improvement in blood tests like cholesterol.

1) Leptin A-200 injections daily with 2 inactive pills taken three times a day, 2) Caffeine with ephedrine pills taken 3 times a day with an inactive injection daily and 3) Both Leptin A-200 injections daily and caffeine with ephedrine pills taken three times a day.

ELIGIBILITY:
Inclusion Criteria:

* You are healthy.
* You are not pregnant or nursing.
* You are between 18 and 60 years of age.
* You have a body mass index, calculated from your height and weight, of 30 to 40 kg/m2.

Exclusion Criteria:

* You take chronic medications except hormone replacement or contraception.
* You are a woman and are unwilling to use effective contraception during the trial.
* You have blood pressure higher than 150/90.
* You have heart disease.
* You have urinary symptoms from an enlarged prostate.
* You have gained or lost more than 10 pounds in the last 6 months.
* You have used a monoamine oxidase inhibitor medication in the last month.
* You have high or low thyroid function that has not been controlled in the normal range for at least 2 months.
* You have heart disease or a history of stroke.
* You have a known sensitivity to E. coli or E. coli derived products.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2001-02; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Compare the percent loss of total body fat to the percent loss of visceral fat with leptin alone, caffeine and ephedrine and the combination of leptin,caffeine and ephedrine. | 28 weeks

SECONDARY OUTCOMES:
Compare the loss of fat and lean tissue with leptin alone. | 28 Weeks
To compare the loss of fat and lean tissue with caffeine with ephedrine alone. | 28 Weeks
compare the loss of fat and lean tissue with leptin, ephedrine and caffeine combination. | 28 Weeks
To compare weight loss with leptin alone. | 28 Weeks
To compare weight loss caffeine with ephedrine alone. | 28 Weeks
To compare weight loss with leptin, ephedrine and caffeine combination. | 28 Weeks
To compare the changes in insulin, with leptin alone. | 28 Weeks
To compare the changes in insulin, with caffeine with ephedrine alone | 28 Weeks
To compare the changes in insulin, with leptin , ephedrine and caffeine combination. | 28 Weeks
To compare the changes in triglycerides, with leptin alone. | 28 Weeks
To compare the changes in triglycerides, caffeine with ephedrine alone. | 28 Weeks
To compare the changes in triglycerides, with leptin , ephedrine and caffeine combination | 28 Weeks
To compare the changes in cholesterol, with leptin alone. | 28 Weeks
To compare the changes in cholesterol, caffeine with ephedrine alone. | 28 Weeks
To compare the changes in cholesterol with leptin , ephedrine and caffeine combination | 28 Weeks
To compare the changes in HDL cholesterol, with leptin alone. | 28 Weeks
To compare the changes in HDL cholesterol, caffeine with ephedrine alone. | 28 Weeks
To compare the changes in HDL cholesterol, with leptin , ephedrine and caffeine combination | 28 Weeks
To compare the changes in LDL cholesterol, with leptin alone. | 28 Weeks
To compare the changes in LDL cholesterol, caffeine with ephedrine alone. | 28 Weeks
To compare the changes in LDL cholesterol, with leptin , ephedrine and caffeine combination | 28 Weeks
To compare the changes in glucose, with leptin alone. | 28 Weeks
To compare the changes in glucose, caffeine with ephedrine alone. | 28 Weeks
To compare the changes in glucose, with leptin , ephedrine and caffeine combination | 28 Weeks
To compare the changes in uric acid, with leptin alone. | 28 Weeks
To compare the changes in uric acid, caffeine with ephedrine alone. | 28 Weeks
To compare the changes in uric acid, with leptin , ephedrine and caffeine combination | 28 Weeks
To compare the changes in Alanine Aminotransferase (ALT )with leptin alone. | 28 Weeks
To compare the changes in Alanine Aminotransferase (ALT ) caffeine with ephedrine alone. | 28 Weeks
To compare the changes in Alanine Aminotransferase (ALT ) with leptin , ephedrine and caffeine combination | 28 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Liu AG, Smith SR, Fujioka K, Greenway FL. The effect of leptin, caffeine/ephedrine, and their combination upon visceral fat mass and weight loss. Obesity (Silver Spring). 2013 Oct;21(10):1991-6. doi: 10.1002/oby.20416. Epub 2013 Jun 11. PMID 23686786